CLINICAL TRIAL: NCT03419767
Title: The Problem of Insulin Resistance in Patients After Carotid Revascularization
Brief Title: Insulin Resistance in Patients After Carotid Revascularization
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZS-1468
Record Dates: First submitted 2018-01-27; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Carotid Stenosis
Keywords: carotid stenosis; melatonin; insulin resistance; inflammation; carotid revascularization; antioxidants
MeSH Terms: conditions — Carotid Stenosis; Insulin Resistance; Inflammation | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgery with melatonin (Active Comparator): Patients under carotid revascularization surgery with melatonin taken during perioperative period.
  Interventions: Drug: Melatonin
- surgery with blank control (Sham Comparator): Patients under carotid revascularization surgery with nothing unnecessary taken during perioperative period
  Interventions: Other: blank

INTERVENTIONS:
Drug: Melatonin — Patients under carotid revascularization surgery taking 6mg/day melatonin orally from 3 days before operation to 3 days after operation.
  Arms: surgery with melatonin
Other: blank — Patients under carotid revascularization surgery without taking melatonin
  Arms: surgery with blank control

SUMMARY:
The main purpose of this study is to study the phenomenon of insulin resistance in patients after carotid revascularization surgery through population-based, randomized, double-blind, placebo-controlled trial.

DETAILED DESCRIPTION:
Trial Title: Insulin Resistance in Patients After Carotid Revascularization. Protocol: Investigators recruited eligible Han Chinese participants (aged 40-80) who were diagnosed with carotid stenosis and had indications for carotid revascularization surgery. Participants were excluded if participants had undergone surgical contraindication, or psychiatric disorders, or cancer, or pregnant, or lactating, or taking antipsychotic drugs during perioperative period. Participants were randomly divided into groups of oral melatonin, and blank control. Participants in groups of oral melatonin took melatonin orally 6mg/day from 3 days before operation to 3 days after operation. Blood samples (about 6 milliliter) were taken at baseline, the first, the second, and the third morning after the operation, all in the fasting state. Through a series hospital clinical laboratory and related ELISA kits to detect the insulin, C-peptide and glucose in serum. Superoxide dismutase (SOD), malonaldehyde (MDA), catalase(CAT), endothelial nitric oxide synthase (eNOS), Interleukin 6 (IL-6), tumour necrosis factor(TNF-α), were included for analysis to verify whether melatonin have protective effect for inflammation and oxidative stress in patients under carotid revascularization, which might be the mechanism of insulin resistance after surgery. This trial is approved by the Ethics Committee of Peking Union Medical College Hospital (No. ZS-1468). All participants completed a questionnaire and signed an informed consent document. Otherwise, participants will get appropriate economic compensation. Trial associates monitored compliance with the masking procedure throughout the trial. All participants and study investigators were unaware of treatment allocation throughout the study. The randomization codes remained sealed until after data collection and cleaning, and completion of a masked analysis. The study team monitored and classified protocol deviations. Investigators summarized baseline clinical and demographic characteristics with descriptive statistics and then determined by the Univariate Analysis of Variance. All the data analyses were done using statistical software SPSS 20.0.

Expected results: Postoperative levels of insulin resistance in both groups are higher than the preoperative. Compared with the blank control group, patients taking melatonin might have lower postoperative levels of insulin resistance, inflammation and oxidative stress.

Consent document: The potential risk, research as a treatment drug of melatonin may delay the metabolism of antipsychotic antipsychotic drug, so when investigators recruit psychiatric disorders or taking antipsychotic drugs orally during the 2 weeks of the trial should exclusion. As a Health care medicine, Melatonin is not suitable for children, so investigators selected recruiting participants under the age of 40 to 80.

The measure to minimize the risk, fully inform the participants and their families the trial's advantages, disadvantages and desired effect. All participants totally agree with the subjects. In this process, at least three or more effective way to get contact with the medical staff or doctor and ensure that those unexpected accident should deserve effective tackle. Participants guarantee to comply with the criterion before start of the trial. Our research involves the application of melatonin is through the china food and drug administration (CFDA) approved to ensure its safety (include its chemical composition, structure, content parameters, main raw material and appropriate crowd). All staff is qualified medical professionals to guarantee the safety of all participants.

The potential risks or discomfort, or inconvenience, or benefits for participants: So far, effective of melatonin in human include regulating sleep, anti-tumor, immune regulation, regulating of inflammation and immune and regulating blood lipid metabolism is confirmed. Adverse reactions is the delay of antipsychotic drug metabolism (so nearly one month ago and during period of the trial participants should not taking antipsychotic drugs) during the trial. The basic principle during the trial is ensure safety of participants.

The relevant content consultation: Everyone have the right to consultation the research content through telephone: +86 01069152500 (principal investigator) and +86 01069155817(Ethics committee).

The rights of withdrew from the trial: Participate in the trial is completely voluntary. If for any reason, participants not willing to participate in, or do not wish to continue to participate in this trial, will not affect the rights and interests of participants. In addition, participants have the right to withdraw this trial at any time. If participants do not accord to the doctor instructions, or for the sake of patients' health and benefits, the doctor or the researchers may also require participants to quit the trial.

The compensation of research: If the participants have any unexpected accident relation with the trial, the compensation and responsibility will be provided by Peking Union Medical College Hospital.

Privacy protection: The privacy of every participant will be protected. The results of the trial in academic publications will not leak any information to identify your personal identity. Peking Union Medical College Hospital will save everybody's data and guarantee not leak without authorization.

Investigators declare no competing interests.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with carotid stenosis
* had indications for carotid revascularization

Exclusion Criteria:

* surgical contraindication
* cardiovascular disease
* psychiatric disorders
* cancer
* pregnant
* lactating
* taking antipsychotic drugs during perioperative period
* history of trauma during perioperative period

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
insulin resistance in patients under carotid revascularization assessed by the concentration of insulin | 3 months
  perioperative insulin resistance detected by the concentration of insulin by ELISA kit
inflammation in patients under carotid revascularization assessed by the concentration of IL-6 | 3 months
  inflammation detected by the concentration of IL-6 by ELISA kit
inflammation in patients under carotid revascularization assessed by the concentration of TNF-α | 3 months
  inflammation detected by the concentration of TNF-α by ELISA kit
inflammation in patients under carotid revascularization assessed by the concentration of eNOS | 3 months
  inflammation detected by the concentration of eNOS by ELISA kit
oxidative stress in patients under carotid revascularization assessed by the concentration of CAT | 3 months
  oxidative stress detected by the concentration of CAT by ELISA kit
oxidative stress in patients under carotid revascularization assessed by the concentration of MDA | 3 months
  oxidative stress detected by the concentration of MDA by ELISA kit
oxidative stress in patients under carotid revascularization assessed by the concentration of SOD | 3 months
  oxidative stress detected by the concentration of SOD by ELISA kit

CONTACTS AND LOCATIONS:
Overall Officials: Changwei Liu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jovanovski-Srceva M, Kuzmanovska B, Mojsova M, Kartalov A, Shosholcheva M, Temelkovska-Stevanoska M, Gavrilovska A, Stavridis S, Spirovski Z, Kondov B, Kokareva A, Todorov R, Spirovska T. Insulin Resistance, Glycemia and Cortisol Levels in Surgical Patients who Had Preoperative Caloric Load with Amino Acids. Pril (Makedon Akad Nauk Umet Odd Med Nauki). 2015;36(3):61-70. doi: 10.1515/prilozi-2015-0079. PMID 27442397
- [Background] de Luis D, Izaola O, de la Fuente B, Aller R. Effect of L-arginine supplementation on insulin resistance and adipocitokines levels in head and neck cancer non diabetic patients after surgery. Nutr Hosp. 2014 Oct 10;30(4):870-5. doi: 10.3305/nh.2014.30.4.7864. PMID 25335675
- [Background] van Stijn MFM, Soeters MR, van Leeuwen PAM, Schreurs WH, Schoorl MG, Twisk JWR, De Bandt JP, Bonnefont-Rousselot D, Cynober L, Ackermans MT, Serlie MJ, Houdijk APJ. Effects of a Carbohydrate-, Glutamine-, and Antioxidant-Enriched Oral Nutrition Supplement on Major Surgery-Induced Insulin Resistance: A Randomized Pilot Study. JPEN J Parenter Enteral Nutr. 2018 May;42(4):719-729. doi: 10.1177/0148607117711691. Epub 2017 Dec 20. PMID 28541810
- [Background] Singh M, Chaudhary M, Vashistha A, Kaur G. Evaluation of effects of a preoperative 2-hour fast with glutamine and carbohydrate rich drink on insulin resistance in maxillofacial surgery. J Oral Biol Craniofac Res. 2015 Jan-Apr;5(1):34-9. doi: 10.1016/j.jobcr.2015.02.006. Epub 2015 Mar 4. PMID 25853046
- [Background] Thorell A, Nygren J, Ljungqvist O. Insulin resistance: a marker of surgical stress. Curr Opin Clin Nutr Metab Care. 1999 Jan;2(1):69-78. doi: 10.1097/00075197-199901000-00012. PMID 10453333
- [Background] Ljungqvist O. Jonathan E. Rhoads lecture 2011: Insulin resistance and enhanced recovery after surgery. JPEN J Parenter Enteral Nutr. 2012 Jul;36(4):389-98. doi: 10.1177/0148607112445580. Epub 2012 May 10. PMID 22577121
- [Background] Zareba K, Kamocki Z, Kuklinski A, Kedra B. Problem of the insulin resistance in surgery. Pol Przegl Chir. 2011 May;83(5):287-91. doi: 10.2478/v10035-011-0045-1. No abstract available. PMID 22166483
- [Background] Wang ZG, Wang Q, Wang WJ, Qin HL. Randomized clinical trial to compare the effects of preoperative oral carbohydrate versus placebo on insulin resistance after colorectal surgery. Br J Surg. 2010 Mar;97(3):317-27. doi: 10.1002/bjs.6963. PMID 20101593
- [Background] Kucukakin B, Gogenur I, Reiter RJ, Rosenberg J. Oxidative stress in relation to surgery: is there a role for the antioxidant melatonin? J Surg Res. 2009 Apr;152(2):338-47. doi: 10.1016/j.jss.2007.12.753. Epub 2008 Jan 10. PMID 18262562
- [Background] Kucukakin B, Lykkesfeldt J, Nielsen HJ, Reiter RJ, Rosenberg J, Gogenur I. Utility of melatonin to treat surgical stress after major vascular surgery--a safety study. J Pineal Res. 2008 May;44(4):426-31. doi: 10.1111/j.1600-079X.2007.00545.x. Epub 2008 Jan 15. PMID 18205732
- [Background] Tangvarasittichai S. Oxidative stress, insulin resistance, dyslipidemia and type 2 diabetes mellitus. World J Diabetes. 2015 Apr 15;6(3):456-80. doi: 10.4239/wjd.v6.i3.456. PMID 25897356
- [Background] Keane KN, Cruzat VF, Carlessi R, de Bittencourt PI Jr, Newsholme P. Molecular Events Linking Oxidative Stress and Inflammation to Insulin Resistance and beta-Cell Dysfunction. Oxid Med Cell Longev. 2015;2015:181643. doi: 10.1155/2015/181643. Epub 2015 Jul 14. PMID 26257839